CLINICAL TRIAL: NCT05372458
Title: The Mechanism Study of Diabetic Pancreatic Amyloid Deposition on Cognitive
Brief Title: The Mechanism Study of Diabetic Pancreatic Amyloid Deposition on Cognitive Dysfunction in Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, YiHui Guan, Professor, Huashan Hospital
Other Study IDs: KY2021-007
Record Dates: First submitted 2022-05-08; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: AD; DM; PET-CT

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alzheimer's disease (AD) is closely related to diabetes (DM). DM will aggravate the progression of AD, but the specific mechanism has not yet been clarified. Previous study found that a key pathological feature of the pancreas in patients with DM is islet amyloid polypeptide, and there is also islet amyloid polypeptide in the brain. Therefore, DM may cause cytotoxicity through the interaction between pancreatic amyloid and brain Aβ protein and further aggravate AD progress. In this study, starting with DM and AD pathological biomarkers, the amyloid PET target molecular probe 18F-AV45 will be used to monitor the dynamic changes of amyloid protein in the brain and pancreas during the development of AD. The completion of this study will provide a new view for understanding the mechanism of DM on AD cognitive dysfunction and effectively preventing and treating these two diseases.

DETAILED DESCRIPTION:
This is a single-center, prospective, and observational study, which mainly focuses on the interaction between pancreatic amyloid and brain Aβ protein and further aggravates AD progress in China. PET imaging will be used on subjects. Previously collected patient data may also be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Non-disease controls:

  1. Age between 60 and 80 years old; gender is not limited.
  2. The investigators have normal cognition and negative Aβ imaging through the test.
  3. Informed consent must be signed in writing by the subjects or their legal guardians and caregivers.
  4. Blood routine: white blood cell count (WBC) 4~10×109/L; platelet (PLT) 100~300×109/L; hemoglobin (HB) 120~160 g/L; renal function: serum creatinine less than or equal to Upper limit of normal range; liver function: bilirubin, AST (SGOT)/ALT (SGPT) less than or equal to the upper limit of normal range; electrocardiogram: no significant abnormality.
  5. Willingness and ability to cooperate with all projects of this research.

AD patients/DM patients:

1. Age between 60 and 80 years old; gender is not limited.
2. The diagnosis of AD was based on the 2011 National Association on Aging and Alzheimer's Disease (NIA-AA) diagnostic criteria for possible AD dementia. The diagnostic criteria for diabetes were based on the 1999 World Health Organization (WHO) diagnostic criteria for diabetes.
3. Brain MRI supports the diagnosis of AD, and there is no evidence of other neurological diseases.
4. No neurological disease, major chronic disease, malignant tumor or acute infectious disease has been confirmed by the investigator.
5. An informed consent form must be signed in writing by the subjects or their legal guardians and caregivers.
6. Blood routine: white blood cell count (WBC) 4~10×109/L; platelet (PLT) 100~300×109/L; hemoglobin (HB) 120~160 g/L; renal function: serum creatinine less than or equal to Upper limit of normal range; function: bilirubin, AST (SGOT)/ALT (SGPT) less than or equal to the upper limit of normal range; electrocardiogram: no significant abnormality.
7. Willingness and ability to cooperate with all projects of this research.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:

  1. Suffering from other serious neurological diseases, or gastrointestinal, cardiovascular, liver, kidney, blood system, tumor endocrine, respiratory system, immune deficiency and other serious diseases.
  2. Candidate subjects have contraindications to PET/CT scanning. Those who cannot accept repeated intravenous injections; those who may be allergic to drugs and their components (including a history of severe allergy or allergic reactions, especially those who are allergic to the tested drugs); phobia of tightness.
  3. In the past year, in addition to participating in the expected radiation exposure of this clinical study, have participated in other research programs or clinical care, resulting in radiation exposure exceeding the effective dose of 50 mSv.
  4. Drug or alcohol abuse for at least 1 month.
  5. The venous condition is poor and cannot tolerate repeated venipuncture.
  6. The candidate subject has received major surgery within the past 3 months; received experimental drug or device treatment (with unclear effect or safety) within 1 month
  7. The candidate subjects have any clinical conditions that the host of this study believes that this preparation may cause or have potential harm.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: clinical or community
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete PET imaging | 50mins from time of injection
  Assessment of PET/CT imaging to detect abeta in patients with AD and DM

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China